CLINICAL TRIAL: NCT07054489
Title: Using Polygenic Scores to Guide Beta-blocker Therapy for Heart Failure With Mildly Reduced Ejection Fraction
Brief Title: UPBEAT: Using Polygenic Scores to Guide BB Therapy in HF With Mildly Reduced EF
Acronym: UPBEAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Lanfear (Other)
Responsible Party: Sponsor-Investigator, David Lanfear, Senior Staff Physician, Henry Ford Health System
Organization: Henry Ford Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17427
Record Dates: First submitted 2025-03-24; First posted 2025-07-08 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure; Polygenic Score
Keywords: Beta blocker; Metoprolol
MeSH Terms: conditions — Heart Failure | interventions — Adrenergic beta-Antagonists

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, two parallel group clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta Blocker (Experimental): This group will be dispensed and titrated on beta blocker according to study protocol.
  Interventions: Other: Beta blocker
- Placebo (No Intervention): This group will be dispensed and titrated on placebo according to study protocol.

INTERVENTIONS:
Other: Beta blocker — Participants randomized to intervention will be dosed and titrated on beta blocker according to study protocol.
  Arms: Beta Blocker

SUMMARY:
This study will use polygenic scores, a tool which describes differences in genetics, to examine effectiveness of beta blocker medication in heart failure patients with ejection fraction of 41-50 percent. The study will also assess beta blockers' effect on the changes in left ventricular end-systolic volume index by MRI.

DETAILED DESCRIPTION:
Heart failure (HF) is a major public health problem that displays wide variation in progression and response to therapy. Beta-blockers (BB) are the cornerstone of treatment for HF reduced ejection fraction (HFrEF) but only ~25% of patients experience a marked and sustained ejection fraction (EF) response, and they can have unwanted side effects (fatigue, depression, erectile dysfunction, others). The potential for Precision Medicine to improve HF care is great, but despite proof of concept, actionable ways are still lacking to use genomic or biomarker strategies to predict response to typical treatment. An important limitation of pharmacogenetics to date is that most studies used candidate gene approaches, assuming other loci are not meaningful. Unbiased approaches (e.g. genome-wide [GW] association) overcome this, but the typical analysis requires stringent significance levels which result in missing potentially important sources of variation. Common complex disease and drug responses are unlikely to be under strong single-loci influence (e.g., Mendelian disease), and instead are likely influenced by many loci that have relatively weak effects (i.e., polygenicity); such phenotypes are better tackled with approaches like polygenic risk scores. The PI has developed and validated a polygenic score for BB drug-response (in terms of mortality benefit) in HF for European ancestry patients and is currently developing a new score for diverse ancestries, particular African ancestry and admixed populations. To move this new paradigm for precision medicine forward to clinical utility, a randomized trial of BB by genomic (polygenic score) subgroups is needed. Moreover, pivotal trials of BB in HF excluded patients with mildly reduced EF (HFmEF, 40-50%), representing a public health issue of significant size (an estimated prevalence of 1.6M Americans) where currently BB may or may not be used and with limited data to guide who should or should not receive this key therapy. HFmEF patients have abnormal systolic function, high event rates, share many characteristics with HFrEF, and the polygenic response score correctly differentiates responders from non-responders in this group, making them the ideal group of patients in which to test genomically targeted BB treatment in a clinical trial. This pilot study will demonstrate feasibility of a future phase 2 study. That study, if successful would potentially revolutionize HF care by demonstrating signs of efficacy in terms of polygenic drug targeting.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89 years
* Ejection Fraction (EF) >40% and =<50% by any modality within 1 year (must be most recent)
* Clinical diagnosis of HF within 1 year, evidenced by any one: Hospital discharge with primary or secondary HF diagnosis, ER discharge with primary diagnosis of HF, ambulatory diagnostic code for HF and diuretic use, BNP>35 ng/L or NTproBNP >125 ng/L at any time

Exclusion Criteria:

* Unable to provide informed consent
* Previous documented EF =< 35%
* Currently on BB >25% target dose
* Uncontrolled hypertension (systolic BP > 180 at enrollment)
* Has contraindications to all BB or intolerance to metoprolol
* Systolic BP < 100 or heart rate <70
* Current cancer requiring active treatment
* Heart transplant or LVAD or expected in the next year
* Life expectancy < 1 year for any reason
* Dialysis dependence or ESRD
* MI/ PCI/ CABG within 90 days prior to enrollment or planned in the future
* Absolute indication for BB other than heart failure (e.g. tachyarrhythmia required BB for rate control, angina)
* If PI decides for any reason participation in trial is not in best interest of the patient

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricle end systolic volume index | Within 6 months of randomization
  LVESVi, measured in mL per square meter; assessed by cardiac MRI

SECONDARY OUTCOMES:
Other MRI ventricular performance characteristics: Left ventricular EF | Baseline and within 6 months of randomization
  Left ventricular EF, measured in percentage
Other MRI ventricular performance characteristics: Left ventricular end-diastolic volume index | Baseline and within 6 months of randomization
  Left ventricular end-diastolic volume index (LVEDVi) as assessed by cardiac MRI, measured in mL per square meter
Clinical effects: blood pressure | Baseline through exit visit, an interval of approximately 6 months
  Change in Blood pressure, measured in mmHg
Clinical effects: Heart rate | Baseline through exit visit, an interval of approximately 6 months
  Change in Heart rate, measured in beats per minute
Change in NT-proBNP levels | Baseline and within 6 months of randomization
  Blood test for biomarker level of N-terminal pro Brain natriuretic protein, measured in ng/L
Quality of life status | Baseline and monthly for duration of approximately 6 months
  Summary score of KCCQ
Functional status | Baseline through exit visit, an interval of approximately 6 months
  Change in 6-minute-walk-test, measured in meters
Clinical safety events | Baseline through 30 days following completion of exit visit
  Measured in all-cause mortality
Clinical safety events | Baseline through 30 days following completion of exit visit
  Measured in heart failure hospitalizations and emergency room visits
Clinical safety events | Baseline through 30 days following completion of exit visit
  Measured in symptomatic hypotension or syncope

CONTACTS AND LOCATIONS:
Overall Officials: David Lanfear, MD, Principal Investigator — Henry Ford Health
Locations (1):
- Henry Ford Health, Detroit, Michigan, United States